CLINICAL TRIAL: NCT00806117
Title: Comparison of Different Adjuvant Treatments Following Radical Surgery in Early Stage Cervical Carcinoma
Brief Title: Comparison of Different Subsequent Treatments After Radical Surgery
Acronym: STARS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Shenzhen People's Hospital (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Department of Gynecologic Oncology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU50102008049
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Concurrent chemoradiation; Randomized controlled clinical trials
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: After radical surgery, eligible patients with risk pathological factors were randomize to three groups.
  Radiotherapy: Group A underwent 50 GY pelvic RT alone. Radiotherapy and drugs: Group B received concurrent weekly cisplatin and RT (CCRT).
  Radiotherapy and drugs: Group C received paclitaxel and bolus cisplatin every three weeks for two cycles before RT, followed by two cycles of chemotherapy (SCRT).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Radiotherapy (RT) (Active Comparator): Radiotherapy
  Interventions: Radiation: Radiotherapy (RT)
- Concurrent chemoirradiation (CCRT) (Experimental): Concurrent chemoirradiation:
  External beam radiation with concurrent weekly platinum chemotherapy
  Interventions: Other: Concurrent chemoirradiation (CCRT)
- Sequence chemo and radiation (SCRT) (Experimental): Sequence chemotherapy and radiotherapy:
  2 cycles chemotherapy of Paclitaxel and Cisplatin before and after the irradiation
  Interventions: Other: Sequence chemotherapy and radiotherapy (SCRT)

INTERVENTIONS:
Radiation: Radiotherapy (RT) — External irradiation 50Gy/5 weeks
  * Lateral: 2 cm lateral to the bony margin of the pelvis
  * Superior: Between L5 and S1
  * Inferior: 2 cm below the obturator foramen Intracavitary boost 30-35Gy/4 weeks(positive vaginal margins only)
  Arms: Radiotherapy (RT)
Other: Concurrent chemoirradiation (CCRT) — Cisplatin 40mg/m2 every week during external irradiation
  Arms: Concurrent chemoirradiation (CCRT)
Other: Sequence chemotherapy and radiotherapy (SCRT) — Paclitaxel 135~175mg/m2 over 3 hours Cisplatin 60~75mg/m2
  Arms: Sequence chemo and radiation (SCRT)

SUMMARY:
Cervical cancer is still the most common gynecologic cancer. There was no obvious increase of the survival over years. The risk of recurrence after radical surgery has increased with positive lymph nodes, positive surgical margins, positive lymphatic vascular space and deep invasion of the cervical stroma. In recent years, the role of chemotherapy for cervical cancer has been gradually recognized. But as a adjuvant therapy post-surgery, if chemotherapy can improve the overall survival rate of patients with adverse pathological prognostic factors is inconclusive.

In this study, in order to investigate the effect and adverse reaction of chemotherapy as the adjuvant therapy post-surgery on patients with adverse pathological prognostic factors, nine hundred and ninety patients will be randomly divided into three groups, comparing radiotherapy alone, concurrent chemoradiation and sequence chemotherapy and radiotherapy (2 cycles chemotherapy of Paclitaxel and Cisplatin before and after the irradiation). The investigators aim to find out the best therapeutic regimen with lowest adverse reaction for cervical cancer with adverse pathological prognostic factors. To guide clinical treatment options.

DETAILED DESCRIPTION:
After radical surgery, patients with stage IB1 to IIA2 cervical cancer who had one or more following pathological factors were recruited: lymph node metastases (LNM), positive parametrium or margins (PPM), lymphatic vascular space involvement (LVSI), deep invasion of cervical stromal (DIS). Eligible patients were randomized to three groups. Group A underwent 50 GY RT alone. Group B received concurrent weekly cisplatin and RT. Group C received paclitaxel and bolus cisplatin every three weeks for two cycles before RT, followed by two cycles.

We have recruited 800 patients till November 2014.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed cervical carcinoma
* Original clinical stage must be Ib~IIa （FIGO）
* Age between 18-65
* With the presence of these four factors after radical surgery:(1)positive lymph nodes,(2)positive parametria, or positive surgical margins,(3)positive lymphatic vascular space,(4)outer one-third invasion of the cervical stroma
* More than 3 months survival is to expect
* Patients must give signed informed consent

Exclusion Criteria:

* The presence of uncontrolled life-threatening illness
* Receiving other ways of anti-cancer therapy
* Residual tumor which can not be removed in the surgery
* Investigator consider the patients can't finish the whole study
* With normal liver function test (ALT、AST>2.5×ULN)
* With normal renal function test (Creatinine>1.5×ULN)
* WBC<4,000/mm3 or PLT<100,000/mm3
* Receive the external pelvic irradiation before the surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Actual)
Dates: Start 2008-02-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 3-Yr
  DFS survival analysis

SECONDARY OUTCOMES:
Overall Survival | 5-Yr
  OS survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph.D., Study Chair — Sun Yat-sen University
Locations (1):
- Department of Gynecologic Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang H, Feng YL, Wan T, Zhang YN, Cao XP, Huang YW, Xiong Y, Huang X, Zheng M, Li YF, Li JD, Chen GD, Li H, Chen YL, Ma LG, Yang HY, Li L, Yao SZ, Ye WJ, Tu H, Huang QD, Liang LZ, Liu FY, Liu Q, Liu JH. Effectiveness of Sequential Chemoradiation vs Concurrent Chemoradiation or Radiation Alone in Adjuvant Treatment After Hysterectomy for Cervical Cancer: The STARS Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Mar 1;7(3):361-369. doi: 10.1001/jamaoncol.2020.7168. PMID 33443541